CLINICAL TRIAL: NCT05613452
Title: Prospective Phase II Clinical Study of Carbon Ion Beam Stereotactic Radiotherapy for Peripheral Type Early-stage Non-small Cell Lung Cancer
Brief Title: Carbon Ion Therapy for Peripheral Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Jian Chen, Clinical Associate Professor, Shanghai Proton and Heavy Ion Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-THLC 2022-03
Record Dates: First submitted 2022-10-26; First posted 2022-11-14 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study arm (Experimental): patients received carbon ion radiotherapy
  Interventions: Radiation: Carbon ion beam radiotherapy

INTERVENTIONS:
Radiation: Carbon ion beam radiotherapy — Patients receive carbon ion radiotherapy of 12GyE per fraction, totally 4 fractions. Patients with tumors ≥4cm should receive at least 4 cycles of platinum-based doublet chemotherapy.

SUMMARY:
To investigate the efficacy of carbon ion therapy for stage Ia-IIa primary peripheral non-small cell lung cancer (NSCLC). The primary endpoint was progression-free survival (PFS), and the secondary endpoint was local control rate, overall survival (OS) and toxicities.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 80.
2. ECOG general status score of 0-2 .
3. Primary non-small cell lung cancer (NSCLC) confirmed by histology or cytological pathology, T1-2N0M0, stage Ia-IIa (AJCC/UICC 8th edition).
4. The location of the tumor belongs to the peripheral type defined in this study (2cm and beyond (≥2cm) from the esophagus, main bronchial tree, spinal cord, heart, great blood vessels, brachial plexus and stomach, and 1cm and beyond (≥1cm) from the chest wall).
5. Medically inoperable, or patient refuses surgery.
6. Adequate organ function: 1). Blood function: absolute neutrophil count (ANC) ≥1.5 x 109/L, platelet count ≥80 x 109/L, hemoglobin ≥9 g/dL 2). Lung function: FEV1>25%, DLCO>25% 3). Cardiac function: no serious pulmonary hypertension, cardiovascular and cerebrovascular diseases, peripheral vascular diseases, serious chronic heart disease and other complications that may affect radiotherapy.4). Adequate liver function: total bilirubin <1.5 times the upper limit of normal value, and AST, ALT<2 times the upper limit of normal value. 5). Adequate renal function: serum creatinine ≤1.5 times the upper limit of normal or calculated creatinine clearance ≥50 ml /min, and urinary protein <2+. Patients with a baseline urinary protein level of 2+ or more should have a 24-hour urine collection and evidence of a 24-hour urinary protein level of 1g or less.
7. Sign the informed consent.

Exclusion Criteria:

1. Multiple primary tumors.
2. Patient fails to comply with the treatment protocol.
3. Complicated with other malignant tumors that have not been controlled.
4. Patient whose particle radiotherapy plan cannot meet the minimum target dose coverage and dose volume limitation requirements, or cannot meet the dose constrains of normal tissue or organs.
5. Chest radiation therapy or radioactive particle implantation history.
6. Cardiac pacemakers or other internal metal prosthesis implants that may be affected by high-energy radiation or may affect the dose distribution to the radiation target area.
7. Pregnancy (confirmed by serum or urine β-HCG test) or lactation period.
8. HIV positive. Hepatitis virus replication phase, need to receive antiviral therapy, but because of concomitant disease cannot receive antiviral therapy. Active stage of syphilis.
9. A history of mental illness may hinder the completion of treatment.
10. With serious comorbidity that may interfere with radiotherapy, including: (a) Acute infectious diseases or acute active phase of chronic infection. b) Unstable angina pectoris, congestive heart failure, myocardial infarction that has been hospitalized in the past 6 months. c) Exacerbations of chronic obstructive pulmonary disease or other respiratory conditions requiring hospitalization. d) Severely impaired immune function. e) Diseases with excessive sensitivity to radiation such as ataxia telangiectasia. f) Other diseases that may affect particle radiotherapy.
11. Other circumstances that the physician considers inappropriate to participate in clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-09-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
disease progression-free survival rate | From date of radiotherapy started until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  disease progression-free survival rate was defined from the start of carbon ion radiotherapy till the date of disease progression at any site or death, or the last follow up.

SECONDARY OUTCOMES:
local control rate | From date of radiotherapy started until the date of first documented local disease progression, assessed up to 100 months
  local control rate was defined was defined from the start of carbon ion radiotherapy till the date of local failure or the last follow-up
overall survival rate | From date of radiotherapy started until the date of death from any cause, assessed up to 100 months
  overall survival rate was defined from the start of carbon ion radiotherapy till the date of death or the last follow-up
Incidence of Treatment-induced Adverse Events [Safety and Tolerability] | From date of radiotherapy started, every 3-4 months within the first 2 years, every 6 months between years 3 and 5, and annually thereafter, assessed up to 100 months
  Treatment-induced toxicities were scored using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03, for events observed after the first dose of irradiation. Toxicities occurred 90 or more days after the completion of CIRT were defined as late toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Jingfang Mao, PHD, Principal Investigator — Shanghai Proton and Heavy Ion Center
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided